CLINICAL TRIAL: NCT02558153
Title: A Randomized Trial of Aperto Paclitaxel Eluting Dilatation Catheter Compared to POBA in Dialysis Fistula
Brief Title: RCT of Paclitaxel DEB Compared to Standard PTA in Dialysis Fistula
Acronym: APERTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groene Hart Ziekenhuis (Other)
Collaborators: Archer Research (Industry)
Responsible Party: Principal Investigator, Dr Peter M.T. Pattynama, MD, PhD. Interventional radiologist, Groene Hart Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL44059.058.13
Record Dates: First submitted 2015-06-07; First posted 2015-09-23 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Complication of Hemodialysis; Vascular Access Complication
Keywords: drug eluting balloon; percutaneous balloon angioplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DEB - drug eluting balloon (APERTO) (Experimental): Percutaneous balloon angioplasty performed with the investigational device, the paclitaxel eluting APERTO balloon
  Interventions: Device: DEB, drug eluting balloon
- standard PTA (Active Comparator): Percutaneous balloon angioplasty performed with the clinical standard, that is, a non-drug-eluting balloon (POBA, plain old balloon angioplasty).
  Interventions: Device: standard PTA

INTERVENTIONS:
Device: DEB, drug eluting balloon — Percutaneous angioplasty performed with a DEB - drug eluting balloon
  Other Names: Paclitaxel eluting balloon
  Arms: DEB - drug eluting balloon (APERTO)
Device: standard PTA — Percutaneous angioplasty performed with a standard balloon
  Other Names: POBA
  Arms: standard PTA

SUMMARY:
A multicenter randomized clinical trial of paclitaxel drug-eluting balloon (DEB) versus standard percutaneous transluminal angioplasty (PTA) to reduce restenosis in 150 patients with haemodialysis access stenoses.

DETAILED DESCRIPTION:
Prospective multicenter randomized (1:1) Investigator Sponsored Trial, in which 150 consecutive patients candidates for percutaneous intervention of haemodialysis access will be randomly assigned to one of two study arms:

1. Treatment Arm: paclitaxel drug-eluting balloon (DEB) dilatation using the APERTO-balloon
2. Control Arm: standard percutaneous transluminal angioplasty (PTA).

The aim is to evaluate the safety and efficacy of paclitaxel drug-eluting balloon (DEB) for the reduction of restenosis in haemodialysis shunts compared to standard percutaneous transluminal angioplasty (PTA).

ELIGIBILITY:
Inclusion Criteria:

All criteria 1-10 must apply for inclusion.

1. Age > 18 years and < 90 years
2. Patient or legally authorized representative providing written informed consent
3. Patient willing and likely to comply with the follow up schedule
4. Patients with previously well functioning hemodialysis access on the arm presenting with any of the following clinical abnormalities as defined in the NKF-DOQI-protocol criteria (National Kidney Foundation 2000):

   * Abnormal physical examination findings (change in bruits, thrill, pulse, etc
   * Abnormal urea recirculation measurements
   * Elevated venous pressure during dialysis
   * Decreased access flow
   * Previous thrombosis in the access line
   * Development of collateral veins
   * Limb swelling
   * Low arterial pressure during dialysis
   * Unexplained decreases in dialysis dose
5. Target Lesion is hemodynamically relevant and consists of MLD ≤ 3 mm. For enrolment this criterium is judged by the local investigator. For final analysis this criterium is based on the result of central reading of the angiogram.
6. Target Lesion(s) is a de-novo or (non-stent) restenosis
7. Target lesion(s) in dialysis fistulas is located at the anastomosis or in the outflow venous trajectory up to the level (but excluding) the subclavian vein
8. Target lesion(s) in dialysis grafts is located at the arterial or venous anastomosis, inside the graft, or in the outflow venous trajectory up to the level (but excluding) the subclavian vein
9. Multiple Target Lesions are allowed per patient which can be treated by a number of APERTO DEB with aggregate max length of 160 mm
10. NON Target Lesions (i.e. in the subclavian vein) must be successfully treated with standard PTA prior to the Target Lesion.

Exclusion Criteria:

None of criteria 1-12 must apply for inclusion.

1. Patients unable to give informed consent
2. Patients enrolled in another study with any investigational drug or device
3. Patients previously enrolled in the APERTO trial.
4. Female patients of child bearing potential without a negative pregnancy test at the time of intervention
5. Major surgical procedures within 30 days prior to this study or planned within 30 days of entry into this study
6. Patients previously treated with a DEB in the hemodialysis access.
7. Patients with a trombosed hemodialysis access.
8. Immature hemodialysis access (unusable due to insufficient shunt flow volume)
9. Lesion treated within 30 days prior to screening
10. Failure to successfully treat non-target lesions prior the Target Lesion
11. In stent restenosis
12. Patients with any known allergy, hypersensitivity or intolerance to ASA, clopidogrel or ticlopidine, paclitaxel, or contrast medium.
13. Graft infection
14. Life expectancy < 1 years

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-06; Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Adequate functioning of the hemodialysis access | 12 months
  Period of adequate functioning of the hemodialysis access after treatment, defined according to the NKF-DOQI protocol criteria

SECONDARY OUTCOMES:
device success | index procedure (day 0)
  ability of the DEB to be delivered, inflated at pressure ≤ RBP, and retrieved from the Target Lesion without burst
Technical Success | index procedure (day 0)
  achievement of a lumen diameter of at least 70% of the nominal diameter of either the DEB or the post dilatation PTA balloon (whichever is bigger) by visual estimate and without bail-out stenting
Clinical Success | 12 months
  improvement in haemodialysis access failure and resumption of normal dialysis for at least one dialysis session after the index procedure
Procedural Success | Index procedure (day 0)
  Technical Success without the occurrence of MAE (MAE defined here as: death, stroke, thrombotic occlusion, allergic reaction, pulmonary events (including pulmonary edema)
MAE - major adverse events | 12 months
  MAE defined as: death or stroke
thrombotic occlusion of target lesion | 12 months
  thrombotic occlusion of target lesion
thrombotic occlusion of target hemodialysis access | 12 months
  thrombotic occlusion of target hemodialysis access
Clinically driven Target Lesion Revascularization (TLR) | 12 months
  Clinically driven Target Lesion Revascularization (TLR)
Clinically driven Target Shunt Revascularization (TSR) | 12 months
  Clinically driven Target Shunt Revascularization (TSR)

CONTACTS AND LOCATIONS:
Overall Officials: Peter MT Pattynama, MD, PhD, Principal Investigator — Groene Hart Ziekenhuis
Locations (10):
- Belgium (2):
  - UZ Leuven, Leuven, Vlaams Brabant
  - ZNA Stuivenberg, Antwerp
- Netherlands (8):
  - Atrium Medisch Centrum. Department of radiology, Heerlen, Limburg
  - Catharina ziekenhuis, Eindhoven, North Brabant
  - St Lucas Andreas Hospital, Amsterdam, North Holland
  - MC Leeuwarden, Leeuwarden, Provincie Friesland
  - Groene Hart Ziekenhuis, Gouda, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - MC Haaglanden, The Hague, South Holland
  - UMC Groningen, Groningen